





Principal Researchers: David González Familiar and Amaia Arregi Agirre

## **INFORMED CONSENT**

| PROJECT TITLE: Elkar Laguntza peer social support program. |
|---|
| lwith |
| DNI declare that I have read the Patient Information Sheet, a copy of which has been given to me. I have received information about the characteristics of the study, as well as the possible benefits and risks that I can expect, the rights that I can exercise, and the provisions on the treatment of data and samples. I have received sufficient information about the study. |
| I know that my identity will be kept secret and that my samples will be identified with a coding system. I am free to revoke my consent at any time and for any reason, without explanation and without adverse effect on any present or future medical treatment. |
| I consent to the use of my samples and associated clinical data as part of this research project. I consent to participate voluntarily. |
| If there is a surplus sample, I affirm that I have been advised of the disposition options at the end of the research project. |
| In this sense: I request the destruction of the surplus sample. I request the incorporation of the surplus sample in the Basque Biobank. |
| Date Patient's signature |
| I confirm that I have explained the characteristics of the research project and the conservation conditions, if applicable, that will be applied to the sample and to the preserved data. |
| Name of the Investigator or the person designated to provide the information: |
| Date Signature |







## CONSENT FOR THE DONATION OF SAMPLES TO THE BASQUE BIOBANK FOR RESEARCH.

| Clinical responsible: | |
|---|---|
| l: | |
| · | ansferring and storing the sample together with |
| the related clinical information to the Basque B | iobank for Research. |
| guarantees of compliance with current legislation | rage, the place of storage, as well as about the on and the possibility of transferring the samples ned that the present consent will be kept in the |
| facilities of the Biobank Node at the Onkologiko | • |
| GIVE my consent for the Onkologikoa Health Codata (except those that identify me) on cancer, | enter to transfer my samples and relevant health |
| give my consent that: | |
| the sample will be used only for projects rel | |
| the sample will be used for any biomedical i | research (preferably related to the disease). |
| I have been advised of the possibility of consent an anonymized form: | ing to donate the sample and associated data in |
| I WISH THE SAMPLES AND DATA TO BE ANC | NYMIZED*. |
| I WISH THE SAMPLES AND DATA TO BE COD | ED**. |
| have been advised of the possibility of receivin | g information regarding my health derived from |
| future genetic analyses that may be performed | on my biological sample (if the sample has been |
| donated in coded form and genetic data have b | een obtained). |
| I request information | |
| I do not want to receive information | |
| Date | Patient's signature |
| to a company that the control of the | and the second s |
| - | es of the storage and security conditions that wil |
| be applied to the sample and to the clinical data | a stored. |
| Name of the responsible clinician | |
| Date | Signature |







- \* coded sample: the sample is identified with a number that only your physician will be able to relate to you.
- \*\* anonymized sample is one that is not associated with identifying data.